CLINICAL TRIAL: NCT03966859
Title: The Effect of Seven-Day Atorvastatin Administration on Emotional Processing, Reward Processing, and Inflammation in Healthy Volunteers
Brief Title: 7-day Atorvastatin and Emotional Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R61966/RE001
Record Dates: First submitted 2019-05-20; First posted 2019-05-29 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Healthy
Keywords: Atorvastatin; Emotional processing; Reward processing; Inflammation (C-Reactive Protein)
MeSH Terms: conditions — Inflammation | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: Participants will be randomised, in a double-blind fashion, to either placebo or atorvastatin. The randomisation code will be drawn up by a researcher not involved in the study using an online randomisation tool (https://www.sealedenvelope.com/simple-randomiser/v1/lists).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The atorvastatin drug and the placebo will be encapsulated in identical capsules. Participants will not be aware of the treatment that they will be receiving; neither will the researcher. Allocation of treatments will be recorded on a Randomisation List, which will be updated when each new participant enters the randomised phase. The list will be held by a scientist uninvolved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive lactose placebo tablets, encapsulated in opaque capsules, and will be asked to take one capsule daily for seven days at night-time, by mouth
  Interventions: Other: Lactose placebo
- Atorvastatin (Experimental): Participants will receive 20mg atorvastatin tablets, encapsulated in opaque capsules, and will be asked to take one capsule daily for seven days at night-time, by mouth
  Interventions: Drug: Atorvastatin 20mg

INTERVENTIONS:
Drug: Atorvastatin 20mg — oral dose, once daily for 7 days
  Other Names: Lipitor; Atorva
  Arms: Atorvastatin
Other: Lactose placebo — oral dose, once daily for 7 days
  Other Names: placebo
  Arms: Placebo

SUMMARY:
Work in our group has revealed that short-term (7-day) administration of antidepressants produces positive biases in the processing of emotional information in healthy volunteers. Such effect might be an important neuropsychological mechanism of antidepressant action.

The current study will investigate the effect of seven-day administration of atorvastatin 20mg on emotional and reward processing tasks in healthy volunteers. There is evidence that statins may exert antidepressant effects via anti-inflammatory and anti-oxidant pathways, and it is therefore predicted that atorvastatin will have positive effects on emotional and reward processing.

DETAILED DESCRIPTION:
Depression is common and associated with considerable health disability. Traditional antidepressants mainly work by modulating monoamine levels in the synaptic cleft; however, the evidence that depression is caused by impaired serotonin or noradrenaline activity is weak and inconsistent, and indeed current antidepressant strategies remain burdened by partial efficacy, poor side-effects profile, and a slow onset of therapeutic action. Therefore, there is a pressing need to develop antidepressant medications with novel non-monoaminergic mechanisms of action - or, conversely, to identify alternative pathophysiological pathways leading to depression that can be targeted with new drugs. Intriguingly, there is growing evidence that both peripheral and central inflammation play a role in the pathophysiology of depression.

Patients with depression consistently show negative biases in emotional processing, which are believed to play a key role in the aetiology and maintenance of their clinical symptoms. Overall, robust evidence suggests that early changes in emotional processing can serve as valid surrogate markers of antidepressant efficacy; for example, seven days' treatment with selective serotonin and noradrenaline reuptake inhibitors (citalopram and reboxetine respectively) compared to placebo decreases the recognition of negative facial expressions and recall of negative versus positive stimuli in healthy volunteers. Conversely, another study using the pro-inflammatory cytokine interferon-α showed that inflammatory-mediated depression can be associated with an increased recognition of negative facial expressions. Furthermore, depression associated with inflammation is characterised by significant symptoms of anhedonia, which has been linked to diminished neural responses to reward anticipation. Such reward-deficit is particularly refractory to conventional serotoninergic and noradrenergic antidepressants, and even the antidepressant bupropion (a noradrenaline and dopamine reuptake inhibitor), whilst inducing positive changes in emotional processing, appears to worsen reward processing. However, the reversal of this deficit in reward processing is still considered as a valuable marker of target engagement for anti-inflammatory drugs in depression, as a more sensitive outcome measure than traditional rating scales designed to capture the global clinical symptomatology.

The 3-hydroxy-3-methylglutaryl-CoA reductase inhibitors or statins are recommended and have been widely used since the '80s for the primary and secondary prevention of cardiovascular diseases. It is now established that these medications have significant anti-inflammatory effects that are independent from their lipid-lowering properties, as well as appearing early in treatment only after seven day of administration. Statins are considered extremely safe drugs: their more common side-effect are muscle pain or weakness (usually mild and quickly responding to stopping or switching medication) and elevation of liver transaminases (significant only in case of pre-existing hepatic disease), whereas more serious adverse events include rhabdomyolysis (very rare but severe myopathy associated with elevated creatine kinase and myoglobinuria), new-onset diabetes mellitus (in predisposed individual with pre-existing hyperglycaemia), and haemorrhagic stroke (in patients with prior haemorrhagic stroke or lacunar infarct); however, clinical trials have ultimately concluded that such adverse events attributed to statin therapy in routine practice are not actually caused by it, especially at doses lower than 80mg/day and when used for less than 52 weeks. Other common (≥ 1/100, < 1/10) but usually mild side-effects include: nasopharyngitis, pharyngo-laryngeal pain, epistaxis, headache, and gastrointestinal disturbances (constipation, diarrhoea, flatulence, dyspepsia, nausea). Importantly, a potential antidepressant effect for statins has been confirmed in animals, as well as clinically in observational and interventional studies. Although their anti-inflammatory and anti-oxidant properties have been involved, the mechanisms underlying the antidepressant effects of statins remain unclear, therefore further translational studies have been advocated in order to elucidate this aspect.

In this exploratory study, we will investigate the effect of seven-day administration of atorvastatin 20mg once daily compared to placebo on emotional and reward processing tasks in 50 healthy volunteers. In view of the previous evidence that statins may exert antidepressant effects via anti-inflammatory and anti-oxidant pathways, we predict that atorvastatin will have positive effect on emotional and reward processing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-50 years
* Sufficiently fluent English to understand and complete the tasks
* Body Mass Index in the range of 18-30
* Participant is willing and able to give informed consent for participation in the study
* Not currently taking any regular medications (except the contraceptive pill)

Exclusion Criteria:

* Currently any regular medications (except the contraceptive pill)
* History or current significant psychiatric illness
* Current alcohol or substance misuse disorder
* History or current significant hepatic disease
* History or current significant neurological condition (e.g. epilepsy)
* Known hypersensitivity to the study drug (i.e. atorvastatin)
* Pregnant, breast feeding, women of child-bearing potential not using appropriate contraceptive measures
* Participation in a study that uses the same or similar computer tasks as those used in the present study
* Participation in a study that involves the use of a medication within the last three months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Accuracy and reaction times during facial expression recognition task | Assessed during the research visit after the seventh day of atorvastatin or placebo administration, i.e. on the eight day after the patient started taking atorvastatin or placebo
  Faces representing varying degrees [from "neutral" (0%) to "full prototypical emotion" (100%) of basic emotions (happiness, fear, anger, disgust, sadness, surprise)] are displayed on the screen and participants are asked to quickly and correctly classify them. Accuracy and reaction times on positive vs negative stimuli are compared between those receiving drug and placebo.
Accuracy and reaction times during faces dot-probe task | Assessed during the research visit after the seventh day of atorvastatin or placebo administration, i.e. on the eight day after the patient started taking atorvastatin or placebo
  Faces acting as positive or negative emotional stimuli (happy or fearful facial expressions) are presented together with a matched neutral face. One is presented above and one below a central fixation point. Subsequently, a probe appears behind one of the two faces and participants are asked to quickly indicate the position of the probe. Accuracy and reaction times on positive vs negative stimuli are compared between those receiving drug and placebo.
Accuracy and reaction times during emotional categorisation task | Assessed during the research visit after the seventh day of atorvastatin or placebo administration, i.e. on the eight day after the patient started taking atorvastatin or placebo
  Words describing positive and negative personality characteristics are presented, and participants are asked to quickly indicate whether they would like or dislike being described with the presented word. Accuracy and reaction times on positive vs negative stimuli are compared between those receiving drug and placebo.
Accuracy during emotional recall task | Assessed during the research visit after the seventh day of atorvastatin or placebo administration, i.e. on the eight day after the patient started taking atorvastatin or placebo
  After a delay from the Emotional categorisation task, participants are asked to recall and write down as many words as possible from it. Accuracy in recall of positive vs negative stimuli are compared between those receiving drug and placebo.
Accuracy and reaction times during emotional recognition memory task | Assessed during the research visit after the seventh day of atorvastatin or placebo administration, i.e. on the eight day after the patient started taking atorvastatin or placebo
  The original personality descriptors in the Emotional categorisation task, plus an equal number of matched distractor words, are presented, and participants are asked to indicate whether they recognise it from the Emotional categorisation task. Accuracy and reaction times on positive vs negative stimuli are compared between those receiving drug and placebo.

SECONDARY OUTCOMES:
Accuracy and reaction times during reward processing | Assessed during the research visit after the seventh day of atorvastatin or placebo administration, i.e. on the eight day after the patient started taking atorvastatin or placebo
  During a computer-based task, participants are instructed to learn and select which images are associated with wins rather than losses. Accuracy and reaction times are assessed and compared between those receiving drug and placebo.
Changes in C-Reactive Protein levels | A blood sample will be drawn on the day of randomisation and on the day of the research visit (i.e. after the seventh day on atorvastatin or placebo)
  Changes in high sensitivity-C Reactive Protein (hs-CRP) from baseline to seven-day, comparing those receiving drug and placebo

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Cowen, MBBS, MD, FRPsych, Principal Investigator — University of Oxford, Medical Sciences Division, Department of Psychiatry
Locations (1):
- Riccardo De Giorgi, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
To comply with the General Data Protection Regulation (GDPR) and the new Data Protection Act, personal data will be deleted as soon as possible after it is no longer needed for the study.
  Screening information: For volunteers who do not wish to be contacted for future studies, screening information (including contact details) will be stored for up to one year of completing study analyses, and then destroyed by shredding. Contact details may be retained after the end of the study for participants who have agreed to be contacted for future studies.
  Consent forms: Consent forms will be kept for 10 years after the end of the study, and then destroyed by shredding.

REFERENCES:
- [Background] Collins R, Reith C, Emberson J, Armitage J, Baigent C, Blackwell L, Blumenthal R, Danesh J, Smith GD, DeMets D, Evans S, Law M, MacMahon S, Martin S, Neal B, Poulter N, Preiss D, Ridker P, Roberts I, Rodgers A, Sandercock P, Schulz K, Sever P, Simes J, Smeeth L, Wald N, Yusuf S, Peto R. Interpretation of the evidence for the efficacy and safety of statin therapy. Lancet. 2016 Nov 19;388(10059):2532-2561. doi: 10.1016/S0140-6736(16)31357-5. Epub 2016 Sep 8. PMID 27616593
- [Background] Cooper CM, et al. Psychological Medicine 2017; Page 1 of 10. doi:10.1017/S00332917170023792017
- [Background] Cowen PJ, Browning M. What has serotonin to do with depression? World Psychiatry. 2015 Jun;14(2):158-60. doi: 10.1002/wps.20229. No abstract available. PMID 26043325
- [Background] Felger JC, Treadway MT. Inflammation Effects on Motivation and Motor Activity: Role of Dopamine. Neuropsychopharmacology. 2017 Jan;42(1):216-241. doi: 10.1038/npp.2016.143. Epub 2016 Aug 2. PMID 27480574
- [Background] Harmer CJ, Shelley NC, Cowen PJ, Goodwin GM. Increased positive versus negative affective perception and memory in healthy volunteers following selective serotonin and norepinephrine reuptake inhibition. Am J Psychiatry. 2004 Jul;161(7):1256-63. doi: 10.1176/appi.ajp.161.7.1256. PMID 15229059
- [Background] Harmer CJ, Duman RS, Cowen PJ. How do antidepressants work? New perspectives for refining future treatment approaches. Lancet Psychiatry. 2017 May;4(5):409-418. doi: 10.1016/S2215-0366(17)30015-9. Epub 2017 Jan 31. PMID 28153641
- [Background] Jain MK, Ridker PM. Anti-inflammatory effects of statins: clinical evidence and basic mechanisms. Nat Rev Drug Discov. 2005 Dec;4(12):977-87. doi: 10.1038/nrd1901. PMID 16341063
- [Background] Jha MK, Trivedi MH. Personalized Antidepressant Selection and Pathway to Novel Treatments: Clinical Utility of Targeting Inflammation. Int J Mol Sci. 2018 Jan 12;19(1):233. doi: 10.3390/ijms19010233. PMID 29329256
- [Background] GBD 2015 DALYs and HALE Collaborators. Global, regional, and national disability-adjusted life-years (DALYs) for 315 diseases and injuries and healthy life expectancy (HALE), 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1603-1658. doi: 10.1016/S0140-6736(16)31460-X. PMID 27733283
- [Background] Kilic FS, Ozatik Y, Kaygisiz B, Baydemir C, Erol K. Acute antidepressant and anxiolytic effects of simvastatin and its mechanisms in rats. Neurosciences (Riyadh). 2012 Jan;17(1):39-43. PMID 22246008
- [Background] Kohler-Forsberg O, Gasse C, Berk M, Ostergaard SD. Do Statins Have Antidepressant Effects? CNS Drugs. 2017 May;31(5):335-343. doi: 10.1007/s40263-017-0422-3. PMID 28303466
- [Background] Li H, Wang C, Zhang S, Sun S, Li R, Zou M, Cheng G. Safety Profile of Atorvastatin 80 mg: A Meta-Analysis of 17 Randomized Controlled Trials in 21,910 Participants. Drug Saf. 2016 May;39(5):409-19. doi: 10.1007/s40264-016-0394-0. PMID 26860922
- [Background] Macin SM, Perna ER, Farias EF, Franciosi V, Cialzeta JR, Brizuela M, Medina F, Tajer C, Doval H, Badaracco R. Atorvastatin has an important acute anti-inflammatory effect in patients with acute coronary syndrome: results of a randomized, double-blind, placebo-controlled study. Am Heart J. 2005 Mar;149(3):451-7. doi: 10.1016/j.ahj.2004.07.041. PMID 15864233
- [Background] McCabe C, Mishor Z, Cowen PJ, Harmer CJ. Diminished neural processing of aversive and rewarding stimuli during selective serotonin reuptake inhibitor treatment. Biol Psychiatry. 2010 Mar 1;67(5):439-45. doi: 10.1016/j.biopsych.2009.11.001. Epub 2009 Dec 24. PMID 20034615
- [Background] Miller AH, Haroon E, Felger JC. Therapeutic Implications of Brain-Immune Interactions: Treatment in Translation. Neuropsychopharmacology. 2017 Jan;42(1):334-359. doi: 10.1038/npp.2016.167. Epub 2016 Aug 24. PMID 27555382
- [Background] NICE. NICE Clinical Guidelines 2014; 181:11. Available from: https://www.ncbi.nlm.nih.gov/books/NBK268908
- [Background] Parsaik AK, Singh B, Murad MH, Singh K, Mascarenhas SS, Williams MD, Lapid MI, Richardson JW, West CP, Rummans TA. Statins use and risk of depression: a systematic review and meta-analysis. J Affect Disord. 2014 May;160:62-7. doi: 10.1016/j.jad.2013.11.026. Epub 2013 Dec 17. PMID 24370264
- [Background] Penn E, Tracy DK. The drugs don't work? antidepressants and the current and future pharmacological management of depression. Ther Adv Psychopharmacol. 2012 Oct;2(5):179-88. doi: 10.1177/2045125312445469. PMID 23983973
- [Background] Roiser JP, Sahakian BJ. Hot and cold cognition in depression. CNS Spectr. 2013 Jun;18(3):139-49. doi: 10.1017/S1092852913000072. Epub 2013 Mar 12. PMID 23481353
- [Background] Walsh AEL, Huneke NTM, Brown R, Browning M, Cowen P, Harmer CJ. A Dissociation of the Acute Effects of Bupropion on Positive Emotional Processing and Reward Processing in Healthy Volunteers. Front Psychiatry. 2018 Oct 16;9:482. doi: 10.3389/fpsyt.2018.00482. eCollection 2018. PMID 30386259
- [Background] Salagre E, Fernandes BS, Dodd S, Brownstein DJ, Berk M. Statins for the treatment of depression: A meta-analysis of randomized, double-blind, placebo-controlled trials. J Affect Disord. 2016 Aug;200:235-42. doi: 10.1016/j.jad.2016.04.047. Epub 2016 Apr 27. PMID 27148902

DOCUMENTS (2):
  • Informed Consent Form (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03966859/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT03966859/Prot_SAP_001.pdf